CLINICAL TRIAL: NCT00003695
Title: A Randomised Trial of Interval Debulking Surgery in Epithelial Ovarian Cancer Suboptimally Debulked at Primary Surgery
Brief Title: Chemotherapy With or Without Surgery in Treating Patients With Stage II or Stage III Ovarian Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066799; MRC-OV06; EU-98063
Record Dates: First submitted 1999-11-01; First posted 2004-03-15 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2007-05

CONDITIONS: Ovarian Cancer
Keywords: stage II ovarian epithelial cancer; stage III ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Drug Therapy; Surgical Procedures, Operative

INTERVENTIONS:
Drug: chemotherapy
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with surgery may kill more tumor cells. It is not yet known whether chemotherapy plus surgery is more effective than chemotherapy alone in treating patients with stage II or stage III ovarian cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy with or without surgery in treating patients with stage II or stage III ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the impact of interval debulking surgery, in terms of survival, disease-free survival, and quality of life, in patients with newly diagnosed stage II or III ovarian cancer and residual macroscopic disease greater than 1 cm after primary surgery.

OUTLINE: This is a randomized study of debulking surgery with concurrent chemotherapy. Patients are randomized to receive chemotherapy alone (arm I) or chemotherapy and interval debulking surgery (arm II). Arm I: Patients receive six courses of platinum-based chemotherapy at intervals of 3 weeks. Arm II: Patients receive three courses of platinum-based chemotherapy at intervals of 3 weeks. In the absence of disease progression, patients undergo interval debulking surgery approximately 21 days after initiation of the third course of chemotherapy. Surgery is then immediately followed by three additional courses of platinum-based chemotherapy. Patients are followed at 6 months after randomization, then every 3 months for the remainder of the first 2 years, then every 6 months for the following 3 years, and then annually thereafter. Quality of life is assessed prior to randomization and before the fourth course of chemotherapy, and then at follow-up visits at 6 months and 1, 2, and 3 years.

PROJECTED ACCRUAL: There will be 1,000 patients accrued into this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed newly diagnosed stage II or III ovarian epithelial cancer Must be planning to receive platinum-based chemotherapy Must be fit for interval debulking surgery Residual macroscopic disease with longest dimension of largest tumor mass greater than 1 cm in diameter documented at primary surgery or postoperatively by imaging

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No concurrent or prior malignancy likely to interfere with protocol treatments or comparison

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1998-05; Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Jacobs, MD, Study Chair — Elizabeth Garrett Anderson Hospital
Locations (1):
- Saint Bartholomew's Hospital, London, England, United Kingdom